CLINICAL TRIAL: NCT07206862
Title: Clinical Evaluation of the Addition of DEBRICHEM® to the Routine Management of Chronic Diabetic Foot Wounds: an Open-label Randomized Controlled Trial (CHEMfoot Study)
Brief Title: CHEMfoot: DEBRICHEM® in Chronic Diabetic Foot Wounds
Acronym: CHEMfoot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DEBx Medical B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHEMfoot
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Diabetic Foot Ulcer Treatment; Diabetic Foot Wounds
Keywords: chemical debridement; DEBRICHEM; topical desiccating agent; TDA; DFU; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Interventional
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEBRICHEM® + conventional wound care (Experimental): Single topical application of DEBRICHEM® (desiccant gel for chemical debridement) at inclusion, then standard wound dressings and care.
  Interventions: Device: DEBRICHEM®
- Conventional wound care only (No Intervention): Mechanical debridement and wound dressing per standard of care

INTERVENTIONS:
Device: DEBRICHEM® — Single topical application of DEBRICHEM® (desiccant gel for chemical debridement) at inclusion, then standard wound dressings and care.
  Other Names: Topical Desiccating Agent; TDA; DEBRICHEM
  Arms: DEBRICHEM® + conventional wound care

SUMMARY:
This multicenter, randomized controlled trial will evaluate the effectiveness and safety of DEBRICHEM®, a topical desiccant gel, when added to standard care for chronic diabetic foot wounds. Chronic diabetic foot ulcers affect up to 25% of people with diabetes and are associated with high risks of infection, hospitalization, amputation, and mortality. Biofilm formation plays a key role in wound chronicity and delayed healing. DEBRICHEM® is designed to chemically debride wounds by removing biofilm in a single topical application, potentially accelerating the healing process.

A total of 242 adult patients with chronic diabetic foot ulcers (≥4 weeks, 0.5-10 cm²) will be randomized to receive either conventional wound care plus a single application of DEBRICHEM® or conventional wound care alone. The primary endpoint is the proportion of patients achieving complete wound healing at 20 weeks. Secondary outcomes include wound size reduction, infection rates, pain, quality of life, sleep, healthcare resource use, and safety.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are a severe complication of diabetes, affecting approximately 20-25% of patients during their lifetime and preceding up to 80% of lower-limb amputations. Chronic wounds are often associated with biofilm formation, which sustains inflammation, delays healing, and reduces the efficacy of mechanical debridement and systemic treatments. New approaches targeting biofilm could improve wound outcomes.

DEBRICHEM® is a CE-marked (Class IIb) medical device developed by DEBx Medical B.V. It is a red, semi-fluid desiccant gel that rapidly binds water molecules in biological material, thereby disrupting biofilm and necrotic tissue. The gel is applied topically for 60 seconds and then rinsed with saline, replacing conventional mechanical debridement. Previous case series and observational data suggest DEBRICHEM® may accelerate granulation and wound closure. However, no randomized controlled trial has yet demonstrated its clinical benefit in diabetic foot ulcers.

The CHEMfoot study is a prospective, open-label, randomized controlled trial conducted at six centers in France. Adults with type 1 or type 2 diabetes and chronic foot ulcers (≥4 weeks, 0.5-10 cm², Texas grade 0-IIC) will be randomized 1:1 to:

Intervention arm: single topical application of DEBRICHEM® plus standard wound care.

Control arm: standard wound care alone, including mechanical debridement and appropriate dressings.

The primary endpoint is the proportion of patients with complete wound healing at 20 weeks, defined as 100% re-epithelialization, wound closure, and absence of exudate, confirmed by blinded investigators and an independent adjudication committee reviewing photographs.

Secondary outcomes include:

Complete healing at 8 and 12 weeks.

≥50% wound surface reduction at 4, 8, 12, and 20 weeks. Change in wound size over time. Local infection rates. Pain (Visual Analog Scale) before/after debridement and during dressing changes.

Quality of life (EQ-5D-5L, EQ-VAS) and sleep (Epworth Sleepiness Scale). Healthcare utilization (hospitalizations, antibiotic prescriptions). Usability of DEBRICHEM® by healthcare professionals (System Usability Scale). Safety outcomes include the incidence and type of adverse events (AE/SAE) related to DEBRICHEM®, as well as pain levels at predefined time points after application (immediately, 2 hours, 24 hours).

A total of 242 patients (121 per arm) will be enrolled to provide 80% power to detect a 20% absolute difference in healing rates (60% vs. 40%) at 20 weeks, assuming a 20% dropout rate. Randomization will be stratified by center and wound size (0.5-5 cm² vs. >5-10 cm²).

The study duration is 12 months (7 months recruitment, 5 months follow-up). Results will provide high-level evidence on whether DEBRICHEM® offers added value to the standard management of chronic diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* Diabetic foot ulcer (toe, dorsal, plantar, or lateral foot) persisting ≥4 weeks without improvement.
* Requires debridement.
* Wound size 0.5-10 cm².
* Texas classification 0-IIC (controlled neuro-ischemic ulcers, localized infection only).
* HbA1c ≤10% in last 3 months. Peripheral arterial disease controlled, no critical limb ischemia (toe pressure >50 mmHg OR ankle pressure >70 mmHg OR TcPO2 >30 mmHg).

Exclusion Criteria:

* Allergy to DEBRICHEM® components.
* Active malignancy, osteomyelitis, fasciitis, exposed cartilage.
* Revascularization <4 weeks prior.
* Systemic infection.
* Pregnant or breastfeeding women.
* Vulnerable populations under legal protection.
* Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12-23 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete wound healing at 20 weeks | 20 weeks
  100% wound surface closure, complete re-epithelialization, and absence of exudate, confirmed by blinded investigator and adjudication committee review of wound photographs.

SECONDARY OUTCOMES:
wound healing wk 8 | week 8
  Complete wound healing at 8
wound healing week 12 | 12 weeks
  Complete wound healing at 12 weeks.
Proportion of patients with ≥50% wound surface reduction | 20 weeks
  Proportion of patients with ≥50% wound surface reduction at weeks 4,8,12 and 20
wound area change | 20 weeks
  Mean change in wound area (absolute cm² and relative %).
Incidence of wound infection | 20 weeks
  Incidence of wound infection at week 4, 8, 12 and 20
Quality of Iife | 20 weeks
  Health-related quality of life (EQ-5D-5L)
Pain Score | 20 weeks
  Pain scores (Visual Analog Scale) before/after debridement, and during dressing changes.
Sleep quality | 20 weeks
  Sleep quality (Epworth Sleepiness Scale).
health resources | 20 weeks
  Health resource use: hospitalizations, antibiotic prescriptions.
treatment usability | 20 weeks
  Usability of DEBRICHEM® (System Usability Scale questionnaire).
Safety by adverse event monitoring | 20 weeks
  Safety: incidence and nature of adverse events and serious adverse events; pain assessment before, immediately after, 2h, 24h and 20 weeks after DEBRICHEM® application.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Sultan, MD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No